CLINICAL TRIAL: NCT02578043
Title: A Multi Center Double Blind Randomized Placebo Controlled Parallel Group Study Comparing Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75% to Onexton™ Gel and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75% to Onexton™ Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLBG 1508
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clindamycin and BPO Gel 1.2%/3.75% (Experimental): Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75% applied to the face once daily for 84 days.
  Interventions: Drug: Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75%
- Onexton™ Gel (Active Comparator): Onexton™ Gel (Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75%) applied to the face once daily for 84 days.
  Interventions: Drug: Onexton™ Gel
- Placebo (Placebo Comparator): Placebo (vehicle of the test product) applied to the face once daily for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75% — Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75% (Taro Pharmaceuticals Inc.)
  Other Names: Clindamycin, BPO
  Arms: Clindamycin and BPO Gel 1.2%/3.75%
Drug: Onexton™ Gel — Onexton™ Gel (Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75%) (Valeant Pharmaceuticals LLC)
  Other Names: Clindamycin, BPO
  Arms: Onexton™ Gel
Drug: Placebo — Placebo (vehicle of the test product) (Taro Pharmaceuticals Inc.)
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the therapeutic equivalence and safety.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the therapeutic equivalence and safety of the test product Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75% to the reference product Onexton™ Gel (Clindamycin and Benzoyl Peroxide Gel 1.2%/3.75%) in the treatment of acne vulgaris and to demonstrate the superiority of the efficacy of these test and reference products over the placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Must have a minimum ≥ 25 non-inflammatory lesions and ≥ 20 inflammatory lesions and ≤ 2 nodulocystic lesions at baseline on the face.
* Must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning to become pregnant during study participation.
* A history or presence of Crohn's disease, ulcerative colitis, regional enteritis, or antibiotic-associated colitis.
* A history of hypersensitivity or allergy to clindamycin, benzoyl peroxide and/or any of the study medication ingredients and its excipients.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 844 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Demonstration of Bioequivalence | Week 12
  Demonstration of Bioequivalence in percent change in inflammatory and non-inflammatory lesion counts

SECONDARY OUTCOMES:
Clinical response of success | Week 12
  The proportion of subjects with a clinical response of success at week 12 defined as an Investigator's Global Assessment score that is at least 2 grades less than the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No